CLINICAL TRIAL: NCT07205887
Title: A Phase 2 Randomized, Dose-Masked Study of Intravitreal EYE103 in Participants With Neovascular Age-Related Macular Degeneration (NVAMD) or Macular Edema Following Branch Retinal Vein Occlusion (BRVO)
Brief Title: A Dose-masked Study of Intravitreal EYE103 in Participants With NVAMD or Macular Edema Following BRVO
Acronym: Super Tuscan
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EyeBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYE-RES-104
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Neovascular Age-Related Macular Degeneration (NVAMD); Branch Retinal Vein Occlusion (BRVO)
Keywords: Neovascular Age-Related Macular Degeneration; Branch Retinal Vein Occlusion; NVAMD; BRVO
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Treatment Naïve NVAMD - Low Dose EYE103 (Experimental): Treatment Naïve NVAMD Cohort - Low Dose EYE103 (50 μL)
  Interventions: Drug: EYE103
- Treatment Naïve NVAMD - High Dose EYE103 (Experimental): Treatment Naïve NVAMD Cohort - High Dose EYE103 (50 μL)
  Interventions: Drug: EYE103
- IR NVAMD - Low Dose EYE103 (Experimental): Incomplete Responder (IR) NVAMD Cohort - Low Dose EYE103 (50 μL)
  Interventions: Drug: EYE103
- IR NVAMD - High Dose EYE103 (Experimental): Incomplete Responder (IR) NVAMD Cohort - High Dose EYE103 (50 μL)
  Interventions: Drug: EYE103
- IR NVAMD - Low Dose EYE103 in combination with Aflibercept 2.0 mg (Experimental): Incomplete Responder (IR) NVAMD Cohort - Low Dose EYE103 (50 μL) in combination with Aflibercept 2.0 mg
  Interventions: Drug: EYE103; Drug: Aflibercept 2.0 mg
- IR NVAMD - High Dose EYE103 in combination with Aflibercept 2.0 mg (Experimental): Incomplete Responder (IR) NVAMD Cohort - High Dose EYE103 (50 μL) in combination with Aflibercept 2.0 mg
  Interventions: Drug: EYE103; Drug: Aflibercept 2.0 mg
- Treatment Naïve BRVO - Low Dose EYE103 (Experimental): Treatment Naïve BRVO Cohort - Low Dose EYE103 (50 μL)
  Interventions: Drug: EYE103
- Treatment Naïve BRVO - High Dose EYE103 (Experimental): Treatment Naïve BRVO Cohort - High Dose EYE103 (50 μL)
  Interventions: Drug: EYE103

INTERVENTIONS:
Drug: EYE103 — EYE103 is a humanized antibody formulated for intravitreal administration
  Other Names: Restoret
Drug: Aflibercept 2.0 mg — Aflibercept 2.0 mg is a commercially available anti-VEGF treatment formulated for intravitreal administration for use in patients with Neovascular Age-Related Macular Degeneration (NVAMD). Aflibercept 2.0 mg is only administered to 2 cohorts of Incomplete Responders (IR) with NVAMD in combination with Low Dose or High Dose EYE103.
  Arms: IR NVAMD - High Dose EYE103 in combination with Aflibercept 2.0 mg; IR NVAMD - Low Dose EYE103 in combination with Aflibercept 2.0 mg

SUMMARY:
EYE-RES-104 is a randomized, dose-masked study of intravitreal EYE103 in participants with neovascular age-related macular degeneration (NVAMD) or macular edema following branch retinal vein occlusion (BRVO).

The study will consist of 4 patient cohorts, with participants in each cohort randomized (1:1) to either a low dose of EYE103 via IVT or a high dose of EYE103 via IVT. 40 participants will be enrolled in each cohort. Enrollment timing for each cohort will be sequenced into specific arms of the study at the Sponsor's discretion.

All participants in the study will receive a total of 3 injections of EYE103 into the study eye, spaced at 4 weeks apart. All participants will return at designated time points following each injection for safety and efficacy assessments. The Week 12 Visit will serve as the end of study visit for all participants.

DETAILED DESCRIPTION:
EYE-RES-104 is a randomized, dose-masked study of intravitreal EYE103 in participants with neovascular age-related macular degeneration (NVAMD) or macular edema following branch retinal vein occlusion (BRVO).

The study will consist of 4 patient cohorts, with participants in each cohort randomized (1:1) to either a low dose of EYE103 via IVT or a high dose of EYE103 via IVT:

* one cohort of 40 treatment naïve NVAMD participants will be randomized (1:1) to 1 of the 2 doses of EYE103 (as monotherapy),
* one cohort of 40 incomplete responder (IR) NVAMD participants will be randomized (1:1) to 1 of the 2 doses of EYE103 (as monotherapy),
* one cohort of 40 IR NVAMD participants will be randomized (1:1) to 1 of the 2 doses of EYE103, to be administered in combination with aflibercept 2.0 mg
* one cohort of 40 treatment naïve BRVO participants will be randomized (1:1) to 1 of the 2 doses of EYE103 (as monotherapy)

Enrollment timing for each cohort will be sequenced into specific arms of the study at the Sponsor's discretion.

All participants in the study will receive a total of 3 injections of EYE103 into the study eye, spaced at 4 weeks apart. IR NVAMD participants in the combination therapy cohort will also receive an injection of aflibercept 2.0 mg in the study eye on Day 1.

All participants will be assessed for safety and efficacy at injection visits. Treatment naïve NVAMD participants and IR NVAMD participants in the monotherapy cohort will also return 2 weeks after each injection visit for safety and efficacy assessments. Depending on the cohort, participants will be evaluated every 2 weeks or every 4 weeks, including measurement of ETDRS BCVA, examination by slit-lamp biomicroscopy, fundoscopy, and SD-OCT. Among other parameters, SD-OCT will be used to measure central subfield thickness (CST) in microns. The Week 12 Visit will serve as the end of study visit for all participants.

ELIGIBILITY:
Inclusion Criteria:

Key General Inclusion Criteria

* Be willing and able to understand the study procedures and the risks involved and provide written informed consent before the first study-related activity
* Be male or female ≥18 years of age.

Key NVAMD-specific Inclusion Criteria

* Be ≥ 50 years of age
* Have treatment naive subfoveal CNV secondary to AMD or juxtafoveal/extrafoveal CNV with foveal involvement
* For participants who are treatment naïve for NVAMD, the diagnosis must have been made within 21 days prior to the Day 1 study treatment

Key IR NVAMD-specific Inclusion Criteria

* Be ≥ 50 years of age
* Have treatment naive subfoveal CNV secondary to AMD or juxtafoveal/extrafoveal CNV with foveal involvement at initial screening
* For participants who are treatment naïve for NVAMD, the diagnosis must have been made within 21 days prior to the Screening Visit 2

Key BRVO-specific Inclusion Criteria

* Be diagnosed with BRVO in the study eye
* Have a decrease in vision in the study eye determined by the Investigator to be primarily the result of BRVO
* Be treatment naïve with vision loss in the study eye and have center-involving macular edema diagnosed within 9 months of Screening

Exclusion Criteria:

Key General Exclusion Criteria

* Be pregnant or breastfeeding
* History of cataract surgery and/or minimally invasive glaucoma surgery in the study eye within 90 days of Screening
* Have had Yttrium-Aluminum Garnet (YAG) laser capsulotomy in the study eye within 90 days of Screening
* Are currently using drugs with known retinal toxicity (e.g., Hydroxychloroquine, pentosan polysulfate sodium, and amiodarone)

Key NVAMD-specific Exclusion Criteria

* Have had previous thermal subfoveal laser therapy in the study eye
* Have had previous photodynamic therapy with Visudyne in the study eye

Key BRVO-specific Exclusion Criteria

* Have macular edema in the study eye considered to be secondary to a cause other than BRVO (eg, DME, NVAMD, Irvine-Gass syndrome)
* Have active iris or angle neovascularization or neovascular glaucoma in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Best-Corrected Visual Acuity measured using the standardized Early Treatment of Diabetic Retinopathy Study (ETDRS) chart | Week 12
  Change from baseline in Best-Corrected Visual Acuity measured using the standardized Early Treatment of Diabetic Retinopathy Study (ETDRS) chart

SECONDARY OUTCOMES:
Changes in retinal central subfield thickness (CST) based on spectral domain optical coherence tomography (SDOCT) | Duration of the study, through Week 12
  Changes in retinal central subfield thickness (CST) based on spectral domain optical coherence tomography (SDOCT)
Changes in Best-Corrected Visual Acuity (BCVA) measured using the standardized Early Treatment of Diabetic Retinopathy Study (ETDRS) chart | Duration of the study, through Week 12
  Changes in Best-Corrected Visual Acuity (BCVA) measured using the standardized Early Treatment of Diabetic Retinopathy Study (ETDRS) chart

CONTACTS AND LOCATIONS:
Overall Officials: Charles Miller, MD PhD, Study Director — EyeBiotech Ltd.
Locations (49):
- United States (49):
  - Scottsdale, Arizona, Scottsdale, Arizona
  - Scottsdale, AZ, Scottsdale, Arizona
  - Glendale, California, Glendale, California
  - Glendale, CA, Glendale, California
  - Modesto, California, Modesto, California
  - Mountain View, California, Mountain View, California
  - Sacramento, CA, Sacramento, California
  - Sactamento, California, Sacramento, California
  - Sacramento, California, Sacramento, California
  - Santa Ana, California, Santa Ana, California
  - Fort Lauderdale, Florida, Fort Lauderdale, Florida
  - Fort Lauderdale, FL, Fort Lauderdale, Florida
  - Lemont, Illinois, Lemont, Illinois
  - Lemont, IL, Lemont, Illinois
  - Hagerstown, Maryland, Hagerstown, Maryland
  - Hagerstown, MD, Hagerstown, Maryland
  - Madison, Mississippi, Madison, Mississippi
  - Madison, MS, Madison, Mississippi
  - Bloomfield, New Jersey, Bloomfield, New Jersey
  - Bloomfield, NJ, Bloomfield, New Jersey
  - Asheville, North Carolina, Asheville, North Carolina
  - Cary, North Carolina, Cary, North Carolina
  - Wake Forest, NC, Wake Forest, North Carolina
  - Wake Forest, North Carolina, Wake Forest, North Carolina
  - West Columbia, SC, West Columbia, South Carolina
  - West Columbia, South Carolina, West Columbia, South Carolina
  - Germantown, Tennessee, Germantown, Tennessee
  - Knoxville, Tennessee, Knoxville, Tennessee
  - Nashville, Tennessee, Nashville, Tennessee
  - Nashville, TN, Nashville, Tennessee
  - Abilene, Texas, Abilene, Texas
  - Amarillo, Texas, Amarillo, Texas
  - Austin, Texas, Austin, Texas
  - Austin, TX, Austin, Texas
  - Bellaire, Texas, Bellaire, Texas
  - Bellaire, TX, Bellaire, Texas
  - Burleson, Texas, Burleson, Texas
  - Dallas, Texas, Dallas, Texas
  - Dallas, TX, Dallas, Texas
  - Plano, Texas, Plano, Texas
  - Round Rock, TX, Round Rock, Texas
  - Round Rock, Texas, Round Rock, Texas
  - San Antonio, Texas, San Antonio, Texas
  - San Antonio, TX, San Antonio, Texas
  - San Marcos, Texas, San Marcos, Texas
  - The Woodlands, Texas, The Woodlands, Texas
  - The Woodlands, TX, The Woodlands, Texas
  - Willow Park, Texas, Willow Park, Texas
  - West Jordan, Utah, West Jordan, Utah